CLINICAL TRIAL: NCT00898989
Title: Evaluation of Muscle Strength and Inflammatory Response in Patients With Inclusion Body Myositis
Brief Title: Muscle Strength and Inflammatory Response in Patients With Inclusion Body Myositis
Acronym: IBMan
Status: Completed | Type: Observational
Sponsor: Institut de Myologie, France (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Olivier BENVENISTE MD PHD, Assistance Publique - Hôpitaux de Paris
Other Study IDs: 2009-a00055-52
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Inclusion Body Myositis
MeSH Terms: conditions — Myositis, Inclusion Body

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Inclusion Body Myositis
- Control

SUMMARY:
Comparison of a group of 20 IBM patients with 20 controls matched on age, gender and weight.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Written consent

Exclusion Criteria:

* Current infection
* Cancer within 1 year
* Immune deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
muscle strength | 2 evaluations at an interval of 9 months

SECONDARY OUTCOMES:
immune response | 1 measure at inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pitié-Salpêtrière, Paris, France